CLINICAL TRIAL: NCT06484101
Title: Effekten av högintensiv träning på Vita Blodkroppar, Med Speciellt Fokus på Funktion Kopplad Till Att bekämpa Cancerceller
Brief Title: Functional Characterization of CD8+ T Cells After Supramaximal Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helene Rundqvist, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-01066-01
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Exercise Induced CD8+ T Cell Recruitment and Characterization of Function and Phenotype of These Cells
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Healthy human subjects performing 3 x 30 seconds of supramaximal exercise with blood obtained before and up to 60 minutes after the exercise bout
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — 3 x 30 seconds of supramaximal exercise

SUMMARY:
Healthy human subjects perform supramaximal exercise with venous blood samples obtained before and up to 60 minutes after the exercise bout.

DETAILED DESCRIPTION:
Healthy, human subjects perform 3 x 30 seconds of supramaximal exercise. Venous blood samples were obtained before and up to 60 minutes after the exercise bout. The blood was used for absolute count of lymphocytes and monocytes per volume blood, and for isolation of CD8+ T cells. It was also used for blood gas analysis. The CD8+ T cells were characterized using flow cytometry, and then cultured for 7 days with CD8+ activation beads. The cells were counted and analyzed for viability at day4 and day8. RNAseq was performed on CD8+ cells isolated before and directly after exercise. CD8+ T cells from Day 1 pre and post exercise and then after 7 days of culture, were analyzed for IFNgamma release using Elispot, and for cytotoxicity against HEK cancer cells in vitro. Flow cytometry of CD8+ T cells was performed on fresh CD8 T cells pre and post exercise, and then on day4 and day8 after culture. SeaHorse metabolic assay was done on Day1 CD8 T cells obtained pre and post exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be used to physical exercise and be able to perform strenous exercise Be able to attend the experimental procedure for the 90 minute duration of the study

Exclusion Criteria:

* Smoking Pregnant Have any medical condition requiring medical treatment

Ages: 20 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
CD8 T cell absolute nr after exercise | Before, directly after, 60 minutes after exercise
  CD8 nr
CD8 T cell cytotoxicity against cancer cells | Cryopreserved CD8 cells from Day 1 and Day 8 of the experiment, obtained before and after exercise
  CD8 T cell lysis of cancer cells
CD8 T cell pheontype after exercise | Before, directly after, 30 minutes and 60 minutes after exercise
  Flow cytometry analysis of CD8 T cells

CONTACTS AND LOCATIONS:
Overall Officials: Helene Rundqvist, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Sjukhuset Huddinge, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT06484101/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT06484101/SAP_001.pdf
  • Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT06484101/ICF_002.pdf